CLINICAL TRIAL: NCT03218033
Title: Improvement of Medication Adherence in Adolescents With SLE Using Web-based Education With and Without a Social Media Intervention
Brief Title: Use of Social Media to Improve Medication Adherence in Adolescents and Young Adults With Systemic Lupus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Children's Miracle Network (Other); Lupus Foundation of America (Other)
Responsible Party: Principal Investigator, Lisabeth Scalzi, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 038689EP
Record Dates: First submitted 2017-07-05; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Systemic Lupus
Keywords: systemic lupus; self-management; social media
MeSH Terms: interventions — Media Exposure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants visited the Facinglupustogether.com website and participated in consecutive weekly modules for 8 weeks. At the end of each module there were questions pertaining to the subject of each module. The control group answered the questions in provided journals and these were sent back to the investigator. All subjects completed surveys in REDCap prior to the study intervention and again 6 weeks after study completion to assess secondary outcome measures. Medication adherence was assessed by calculating a medication possession ratio by acquiring information on fill dates at the subjects' pharmacies.
- Social Media (SM) (Active Comparator): The intervention phase was 8 weeks in duration. Participants visited the Facinglupustogether.com website and participated in consecutive weekly modules. 8 The SM group answered the questions at the end of each module on a blogging site with other SM participants. SM participants were encouraged to provide feedback or questions about the material or personal questions that arose in response to each module.
  All subjects completed surveys in REDCap prior to the study intervention and again 6 weeks after study completion to assess secondary outcome measures. Medication adherence was assessed by calculating a medication possession ratio by acquiring information on fill dates at the subjects' pharmacies.
  Interventions: Behavioral: Social Media

INTERVENTIONS:
Behavioral: Social Media
  Arms: Social Media (SM)

SUMMARY:
The goal of this study was to examine the effect of an online educational program with and without a social media experience.The primary goal of this study was to determine whether medication adherence would be improved by having adolescents and young adults with systemic lupus erythematosus participate in an online educational website, with or without a social media experience. The secondary goal was to determine whether secondary outcomes such as quality of life, stress, and self-efficacy improved in this model, and whether these changes were associated with improvements in medication management.

DETAILED DESCRIPTION:
Self-management skills, including medication management, are vital to the health of adolescents and young adults with systemic lupus erythematosus (SLE). Non-adherence with medications in patients with systemic lupus has been noted to be as poor as 40%. Success in disease control can be significantly impacted by such non-adherence. Poor medication compliance is associated with higher SLE disease activity scores and higher SLE disease activity in turn has been demonstrated to be significantly associated with a decline in quality of life. Much attention has been paid to how to improve self-management skills in adults, but less is known about how to target adolescents, an age group with a complex set of emotional and developmental needs.

The goal of this study was to examine the effect of an online educational program with and without a social media experience.The primary goal of this study was to determine whether medication adherence would be improved by having adolescents and young adults with SLE participate in an online educational website, with or without a social media experience. The secondary goal was to determine whether secondary outcomes such as quality of life, stress, and self-efficacy improved in this model, and whether these changes were associated with improvements in medication management.

ELIGIBILITY:
Inclusion Criteria:

* age between 13 and 23 at the time of recruitment
* having the diagnosis of SLE made or confirmed by a pediatric or adult rheumatologist at Penn State Children's Hospital/Hershey Medical Center
* having regular internet access.

Exclusion Criteria:

* age <13 or >23 years
* comorbid medical or psychiatric illness that would affect the outcome measures.

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Medication Adherence | 6 months
  A medication possession ratio was calculated based on fill date information from the subjects' pharmacies

SECONDARY OUTCOMES:
Stress utilizing the Perceived Severity of Stress Questionnaire | 14 weeks
  Stress was measured by the Perceived Severity of Stress Questionnaire (PSQ)
Self-efficacy utilizing the Children's Arthritis Self-Efficacy scale | 14 weeks
  Self-efficacy was measured using the Children's Arthritis Self-Efficacy scale (CASE) which was modified slightly for systemic lupus
Quality of Life utilizing the Simple Measure of the Impact of Lupus Erythematosus in Youngsters (SMILEY) index | 14 weeks
  Quality of life was assessed using the validated Simple Measure of the Impact of Lupus Erythematosus in Youngsters (SMILEY) index
Sense of agency | 14 weeks
  Sense of agency (SOA) was measured via three Likert scale questions aimed to tap three core concepts of agency: competence ("Blogging… makes me feel I have control over my own voice"), assertiveness ("…enables me to assert myself"), and confidence ("…makes me feel I have a distinct voice")
Sense of community | 14 weeks
  Sense of community (SOC) was measured using a 22-item scale (8, 9, 20). SOC consists of feelings of belonging to the community, having influence on, and being influenced by, the community, being supported by the community while also supporting them; and feelings of shared emotional connection.
Empowerment | 14 weeks
  Empowerment was assessed using a validated quantitative Likert scale tool that measured 1) "empowering processes" (Appendix A), and 2) "empowering outcomes"

REFERENCES:
- [Derived] Scalzi LV, Hollenbeak CS, Mascuilli E, Olsen N. Improvement of medication adherence in adolescents and young adults with SLE using web-based education with and without a social media intervention, a pilot study. Pediatr Rheumatol Online J. 2018 Mar 14;16(1):18. doi: 10.1186/s12969-018-0232-2. PMID 29540181